CLINICAL TRIAL: NCT02527447
Title: A Pilot Study of Biomarkers for Personalized Early Assessment of Response During Salvage Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Biomarkers for Personalized Early Assessment of Response During Salvage Chemotherapy in People With Relapsed or Refractory Acute Myeloid Leukemia (PEARL15)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150176; 15-H-0176
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10-28

CONDITIONS: Acute Myeloid Leukemia
Keywords: Measurable Residual Disease; Relapsed/Refractory AML; Salvage Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

-Acute myeloid leukemia (AML) is a cancer of the white blood cells. It can be fatal. Standard treatment involves intensive chemotherapy. Not all treatment works. AML that has not responded to treatment (refractory) or that has returned after treatment (relapsed) is high-risk even with treatment. Success of therapy is normally determined after 28 to 56 days. This study will see if a blood test on day 4 of therapy can help identify earlier those who will not respond.

Objectives:

-To see if a blood test on day 4 of therapy can help identify those who will not respond to treatment for AML.

Eligibility:

-People ages 18-70 who have refractory or relapsed AML and have had at least one previous therapy for it.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Participants will have:
* Several blood tests.
* Bone marrow exams: a needle is inserted into the hip to take cells from the bone marrow.
* Echocardiogram: a small probe is held to the chest to take pictures of the heart.
* ECG: soft electrodes are stuck to the skin. A machine records the heart s signals.
* CT scans: they will lie in a machine that takes pictures of the body.
* Standard chemotherapy.
* Possible transfusions of blood products such as red blood cells or platelets.
* Participants will be expected to stay in the study typically for 2 3 months. This will include inpatient treatment. Inpatient stay normally will be 1 or 2 months.

DETAILED DESCRIPTION:
Effective treatment of patients with relapsed and refractory acute myeloid leukemia (RR-AML) remains a significant unmet need. Current response criteria were originally proposed in 1956 and do not provide a sensitive assessment of AML disease burden, as evidenced by the disconnect between the apparent success of current induction therapy in achieving complete remission in most patients and the stark reality of median overall survival times of less than two years. While sensitive minimal/measurable residual disease assays assessing AML disease burden have been developed, the role for these tests in the treatment algorithm for patients with RR-AML has yet to be defined. We propose evaluating if these high sensitivity assays could function as early predictors of salvage therapy failure.

This protocol is designed as a feasibility study to evaluate if use of high sensitivity peripheral blood-based molecular assays on day 4 of induction salvage chemotherapy can predict failure to ultimately achieve a CR or CRi in patients with RR-AML. Eligible patients will receive salvage induction therapy using FDA approved antineoplastic agents given either alone or in combinations as defined in the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for AML.

Additional secondary objectives include investigating the relationship between kinetics of gene expression changes and response to chemotherapy, determining the proportion of patients for whom results of day 4 peripheral blood gene expression testing are available before day 8 of therapy, determining the proportion of patients for whom results from pre-treatment molecular and genetic testing are available before day 8 of therapy, assessing patient and disease specific factors associated with failure to achieve a CR, determining the feasibility of measuring AML residual disease burden using alternative technologies and alternative tissue sources, determining the proportion of patients who receive allogeneic hematopoietic stem cell transplant after completion of therapy, determining the incidence of infectious complications with the use of modern prophylactic antimicrobial agents compared with historical comparisons and determining the feasibility of recruiting patients with RR-AML to the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Unequivocal diagnosis of relapsed or refractory acute myeloid leukemia (AML) according to WHO criteria confirmed by bone marrow evaluation within 30 days prior to study enrollment
* Age 18-70 years inclusive
* ECOG performance status of 0 to 2
* Must have received at least one prior AML therapy before study enrollment
* Ability to comprehend the investigational nature of the study and provide informed consent
* Availability of a physician willing to assume clinical care after completion of this research study.
* Subject agreement to use a medically-approved method of contraception to avoid pregnancy throughout the study if a woman of childbearing potential or a male subject with partner of childbearing potential.

EXCLUSION CRITERIA:

* Diagnosis of acute promyelocytic leukemia
* Decreased oxygen saturation at rest (e.g. pulse oximeter less than 88% or PaO2 less than or equal to 55 millimeters of mercury)
* Clinically significant active infection not responding adequately to therapy
* Known positive or history of HIV; active Hepatitis B or C infection. If unknown, screening will be done but results are not needed before proceeding with treatment
* Prior allogeneic hematopoietic stem cell transplant
* Additional malignancy requiring concurrent treatment
* Uncontrolled hepatic, renal, cardiac, gastrointestinal, pulmonary, neurologic, infectious, metabolic or other disease of such severity, which in the opinion of the PI, would preclude ability to tolerate protocol.
* Severe psychiatric illness or complex social situations that would limit the patient s ability to tolerate and/or comply with study requirements.
* Active central nervous system (CNS) leukemic infiltration
* Current pregnancy or breastfeeding
* Prolonged QTc interval prior to therapy (>470ms)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-18; Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this protocol are the outcomes of the blood test performed on day 4 during chemotherapy, and the standardresponse criteria including morphological bone marrow examination following chemotherapy. | 4 days
  The primary outcome of this protocol are the outcomes of the blood test performed on day 4 during chemotherapy, and the standard response criteria at day 30 including morphological bone marrow examination following chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Hourigan, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States